CLINICAL TRIAL: NCT00270608
Title: How Does Early Age Life Style Affect Bone Strength and General Health at Middle Age? Twenty-Five Year Follow-up Health Status Comparison of a Sedentary Versus Extremely Physically Active Population From an Early Age
Brief Title: How Does Early Age Life Style Affect Bone Strength and General Health Parameters at Middle Age?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 12-17.02.06-HMO-CTIL
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Bone Diseases
Keywords: Hypertension; Peripheral vascular disease; Diabetes; Total body fat percentage
MeSH Terms: conditions — Bone Diseases; Hypertension; Peripheral Vascular Diseases; Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Quantitative Computed Tomography of the tibia and spine — a single time 1 minute procedure
Procedure: MRI of the spine and the right knee — a single time 45 minutes procedure
Procedure: Blood test — A single time procedure to check lipid profile and hemoglobin A1C

SUMMARY:
The purpose of this study is to evaluate the effect of vigorous physical activity versus extremely sedentary life style during young age on the bone mineral density and general health in later life.

DETAILED DESCRIPTION:
Bone strength and peak bone mass are preliminary determined by genetic factors. Life style, especially exercise, is also considered to have an important effect on bone strength. Bone has the ability to strengthen itself according to Wolff's Law. When bone is subjected to strains and/or strain rates higher than the usual, it responds by remodeling, strengthening its architecture. The ability is greatest in young individuals and decreases with age. In the elderly this ability is largely non-existent and bone mass is lost. Whether this loss leads to osteoporosis is largely a function of the peak bone mass achieved before the decline. 11% of males and 44 % of females over 50 suffer from osteoporosis in later life. To what extent vigorous exercising beginning at a young age can increase bone strength is not known.

The purpose of the proposed research is to quantify the effect of life style on bone strength and general health parameters by comparing two male populations, one sedentary and the other that has done demanding physical training: (1) Elite infantry recruits who were inducted into the I.D.F. in Feb 1983, did their basic training at Sanur and were part of the 1983 stress fracture project who completed three years of elite infantry service and continued to serve as combat soldiers in the reserves; (2) Yeshiva students who had profiles of 82 or 97 and received deferment from their military service in 1983 and since then have continued their studies and never served in the army.

50 subjects will be reviewed in each group. Measurements of weight, height, waist and abdominal girth, resting pulse and blood pressure will be made. The brachial/ankle blood pressure index will be recorded. MRI of the right knee to study potential degenerate changes will be done using a 1.5 Tesla General Electric Signa MR scanner. Quantitative Computed Tomography (QCT), one of the most popular and effective methods utilized for osteoporosis screening, will be performed to determine volumetric BMD, BMC, bone geometric properties and strength indexes of the tibia and lumbar spine.

Comparisons:

Group I: 50 males (age 41-45), former elite Israeli infantry soldiers, selected randomly from those recruits who did their infantry basic training at Sanur in Feb. 1983 (all profiled 82 or 97) and completed their military service as combat soldiers will be compared to:

Group II: 50 age-, profile- and ethnically-matched Israeli citizens whose military service was deferred in 1983 because of Torah studies and who did not do army service and were not involved in any kind of physical training.

ELIGIBILITY:
Inclusion Criteria:

* Israeli military profile 82 or 97 at age 17-22

Exclusion Criteria:

* Israeli military profile less than 82 at age 17-22
* Former soldiers with shrapnel injuries will be excluded from MRI studies

Ages: 40 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Israeli males who were 17-22 years-old and received a military profile of either 82 or 97 in 1983
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Charles Milgrom, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Milgrom C, Giladi M, Stein M, Kashtan H, Margulies JY, Chisin R, Steinberg R, Aharonson Z. Stress fractures in military recruits. A prospective study showing an unusually high incidence. J Bone Joint Surg Br. 1985 Nov;67(5):732-5. doi: 10.1302/0301-620X.67B5.4055871.